CLINICAL TRIAL: NCT06154213
Title: Building Habits Together Online Weight Loss Program: Pilot Trial
Brief Title: Building Habits Together Online Weight Loss Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Connecticut (Other)
Collaborators: Worcester Polytechnic Institute (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Sherry Pagoto, Professor, University of Connecticut
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HR22-0155; R34HL145439 (NIH)
Record Dates: First submitted 2023-05-23; First posted 2023-12-04 (Actual); Results first posted 2025-03-30 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Obesity
Keywords: obesity; lifestyle intervention; mobile app
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Building Habits Together (Experimental): The Building Habits Together arm includes the 24-week, Facebook-delivered lifestyle intervention based on the Diabetes Prevention Program and use of the Habit app (temptation tracking, exercise planning, and problem solving features).
  Interventions: Behavioral: Building Habits Together
- Getting Healthy Together (Active Comparator): The Getting Healthy Together arm includes the 24-week, Facebook-delivered lifestyle intervention based on the Diabetes Prevention Program and use of the MyFitnessPal app (daily calorie tracking, exercise tracking).
  Interventions: Behavioral: Getting Healthy Together

INTERVENTIONS:
Behavioral: Building Habits Together — Private, hidden Facebook group "Building Habits Together" includes 24 weeks on content based on the Diabetes Prevention Program and the Habit app.
  Arms: Building Habits Together
Behavioral: Getting Healthy Together — Private, hidden Facebook group "Getting Healthy Together" includes 24 weeks on content based on the Diabetes Prevention Program and the MyFitnessPal app.
  Arms: Getting Healthy Together

SUMMARY:
The purpose of this pilot trial is to evaluate the feasibility of a lifestyle intervention where participants will all receive online weight loss counseling delivered via a private Facebook group, but be randomized to the Habit app (developed by the investigators) or MyFitnessPal, a commercial calorie tracking app.

DETAILED DESCRIPTION:
The purpose of this pilot trial is to evaluate the feasibility of a program where 70 adults with overweight or obesity will receive online weight loss counseling delivered via a private Facebook group, but be randomized to the Habit app (developed by the investigators) or MyFitnessPal, a commercial calorie tracking app. Participants randomized to the Habit app will be asked to record their weight daily, monitor their dietary temptations, plan their exercise, and solve diet and exercise related problems. The temptation tracker helps users identify triggers and track when and why those triggers lead to dietary lapses. The exercise planner allows users to plan their exercise for the week and track whether they completed or missed the exercise and why they missed it. The Habit app provides insights to users about the patterns of their dietary lapses and exercise habits. The problem solver feature helps users identify their biggest problem with diet/exercise and then asks a series of questions to help the app provide tailored solutions to the participant to work on. Participants randomized to MyFitnessPal will track their calorie intake and exercise daily during the intervention.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old
* Body mass index (BMI) 27-45 kg/m2
* Wi-Fi connectivity at home
* Logs into Facebook at least 5 days per week over the past 2 weeks
* Has posted/replied on Facebook at least once a week in the past 2 weeks
* Able to participate in the study in English
* Interested in losing weight

Exclusion Criteria:

* Under the age of 18 and over the age of 65
* BMI under 27 or over 45 at screening; then under 27 at the point of the first weight on scale
* Does not have Wi-Fi connectivity at home
* Does not have a Facebook account
* Does not log into Facebook at least 5 days per week over the past 2 weeks
* Did not post/reply on Facebook once a week over the past 2 weeks
* Not able to participate in the study in English
* Does not live in the United States
* Not interested in losing weight
* Pregnant/lactating or plans to become pregnant during study period
* Reports having bipolar disorder, substance abuse, psychosis, an eating disorder, or severe depression
* Had bariatric surgery or plans to have surgery during the study
* Currently taking medication affecting weight
* Has lost ≥5% of weight in past 3 months
* Is participating or intends to participate in another weight loss program during the study that provides coaching or problem solving
* Chronic pain that interferes with the ability to exercise
* Has Type 1 Diabetes
* Has Type 2 Diabetes
* Unable to make dietary changes or increase physical activity
* Unable to walk ¼ mile unaided without stopping
* Currently smokes or vapes nicotine
* No phone connectivity at home and work
* Has a digestive disorder/condition that precludes dietary changes
* Meets criteria for severe depression on the Patient Health Questionnaire (PHQ)-8 (score of >19)
* Does not currently own a smartphone
* Smartphone type and/or version not meeting app requirements
* Participated in previous weight loss studies under the PI
* Unable to attend the orientation webinar
* If University of Connecticut (UConn) employee/student has concerns about being in a Facebook group with other UConn faculty, staff, and students
* Had major surgery in past 6 months and have not been cleared by their doctor to resume physical activity and diet changes
* Plans to have major surgery in the next 6-months
* Has an implanted cardiac defibrillator or pacemaker
* Did not complete screening and on-board processes of study (screening survey, webinar, e-consent, baseline survey, app set-up, scale set-up, etc.)
* Not willing to be audiotaped for focus groups
* Prisoner; or
* Unable to provide consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2023-04-03 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sherry Pagoto, PhD, Principal Investigator — University of Connecticut
Locations (1):
- University of Connecticut, Storrs, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Building Habits Together | Getting Healthy Together
Started | 35 | 35
Completed | 33 | 35
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Building Habits Together | Getting Healthy Together | Total
Number analyzed (Participants) | 35 | 35 | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.1 (12.0) | 46.4 (11.4) | 44.7 (11.7)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 26 | 25 | 51
  Male | 8 | 9 | 17
  Non-binary | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 2 | 14
  Not Hispanic or Latino | 23 | 33 | 56
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 4 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 13 | 20
  White | 20 | 16 | 36
  More than one race | 4 | 2 | 6
  Unknown or Not Reported | 0 | 0 | 0
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 33.5 (5.1) | 34.4 (5.1) | 33.9 (5.1)

OUTCOME MEASURES:

1. Primary Outcome: Mobile App Use
Description: Investigators will calculate the number of days participants used their assigned app
Time Frame: 24 weeks
Measure: Median (Inter-Quartile Range); unit: days out of 168 total
Arm/Group | Building Habits Together | Getting Healthy Together
Number analyzed (Participants) | 35 | 35
days out of 168 total | 18 [7 to 32] | 33 [10 to 118]

2. Primary Outcome: Retention
Description: Investigators will calculate retention as the proportion of participants who provide weight data at the 24 week follow-up
Time Frame: 24 weeks
Measure: Number; unit: participants
Arm/Group | Building Habits Together | Getting Healthy Together
Number analyzed (Participants) | 35 | 35
participants | 33 | 35

3. Primary Outcome: Engagement Per Participant in the Facebook Group
Description: For each participant, investigators will calculate total engagement in the Facebook group as defined as reactions (e.g., like, care, wow, etc.), replies, posts, and poll votes during the 24-week program. Then we will calculate mean or median engagement per participant over 24 weeks.
Time Frame: 24 weeks
Measure: Median (Inter-Quartile Range); unit: total reactions, replies, posts, votes
Arm/Group | Building Habits Together | Getting Healthy Together
Number analyzed (Participants) | 35 | 35
total reactions, replies, posts, votes | 112 [27 to 251] | 96 [40 to 243]

4. Primary Outcome: Ease of Use (Acceptability)
Description: Participants will rate how easy it was to use their assigned app (% who strongly agree/agree)
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Building Habits Together | Getting Healthy Together
Number analyzed (Participants) | 35 | 35
Participants | 18 | 20

5. Primary Outcome: Contamination
Description: Investigators will report the percent of participants in the Habit condition that used MyFitnessPal or other calorie tracking apps during the program.
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Building Habits Together
Number analyzed (Participants) | 35
Participants | 0

6. Primary Outcome: Time Consuming (Burden)
Description: Participants will rate their assigned app in terms of whether they felt it took too much time out of their day (% who strongly agree/agree)
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Building Habits Together | Getting Healthy Together
Number analyzed (Participants) | 35 | 35
Participants | 6 | 8

7. Secondary Outcome: Percentage of Baseline Weight Lost at 24 Weeks
Description: Investigators will calculate percent weight change from baseline at 24 weeks
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: percent baseline weight lost
Arm/Group | Building Habits Together | Getting Healthy Together
Number analyzed (Participants) | 33 | 35
percent baseline weight lost | 2.1 (5.6) | 5 (5.8)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Building Habits Together | Getting Healthy Together
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/35
Serious Adverse Events (participants affected / at risk) | 1/35 | 0/35
Other Adverse Events (participants affected / at risk) | 0/35 | 0/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Building Habits Together (N=35) | Getting Healthy Together (N=35)
kidney failure (Renal and urinary disorders) | 1 (1) | 0 (0) — Participant was admitted to the hospital following blood work that revealed potential kidney failure stage 4/5.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-01): https://cdn.clinicaltrials.gov/large-docs/13/NCT06154213/Prot_SAP_000.pdf